CLINICAL TRIAL: NCT06577285
Title: The Effect Of Botulinum Toxin A In Patients With Excessive Gingival Display With And Without Zinc And Phytase Supplementation: A Randomized Clinical Trial
Brief Title: The Effect Of Botox In Patients With Gummy Smile With And Without Zinc And Phytase Supplementation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mawda Mohamed Hussain Eltoum, Principle investigator Mawada Mohamed Master Degree Student, Periodontology department, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18514PER3_3_1
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Excessive Gingival Display
Keywords: Botulinum Toxin A; Excessive Gingival Display; Zinc And Phytase Supplementation; Botox Injection; Gummy Smile
MeSH Terms: interventions — gluconic acid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group I (Active Comparator): Patients in the intervention group I will take zinc gluconate 50 mg (Now food company) 1 per day to increase zinc level with phytase supplement 176mg (800FTU) (Goodphyte company) 2 tablets per day to give the maximum absorption of zinc, both supplements will be given for 4 days before botulinum toxin injections.
  Interventions: Dietary Supplement: zinc gluconate 50 mg with phytase supplement 176mg (800FTU)
- Intervention group II (Active Comparator): Patients in the intervention group II will take zinc gluconate 50 mg (Now food company) 1 per day to increase zinc level, 4 days before botulinum toxin injections.
  Interventions: Dietary Supplement: zinc gluconate 50 mg
- Control group (No Intervention): Patients in the control group will receive the Botulinum toxin injections only.

INTERVENTIONS:
Dietary Supplement: zinc gluconate 50 mg with phytase supplement 176mg (800FTU) — zinc gluconate 50 mg1 per day with phytase supplement 176mg (800FTU) (Goodphyte company) 2 tablets per day
  Arms: Intervention group I
Dietary Supplement: zinc gluconate 50 mg — zinc gluconate 50 mg 1 per day, 4 days before botulinum toxin injections.
  Arms: Intervention group II

SUMMARY:
Participants with esthetic concern of excessive gingival display who meets the inclusion criteria, will be carried out including history taking, clinical examination and initial therapy.

The initial therapy will consist of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques. Patients who have inadequate crown length and width ratio or short clinical crown will receive esthetic crown lengthening procedure to adjust gingival levels before being included in this study.

Patients in the intervention group I will take zinc gluconate 50 mg 1 per day to increase zinc level with phytase supplement 176mg (800FTU) 2 tablets per day to give the maximum absorption of zinc, both supplements will be given for 4 days before botulinum toxin injections. Patients in the intervention group II will take zinc gluconate 50 mg 1 per day to increase zinc level, 4 days before botulinum toxin injections.

Patients in the control group will receive the Botulinum toxin injections only Clinical photographs will be taken at baseline, 2 weeks, 1 month, 3 months postoperatively.

DETAILED DESCRIPTION:
Initial examination:

Participants with esthetic concern of excessive gingival display who meets the inclusion criteria, will be carried out including history taking, clinical examination and initial therapy.

The initial therapy will consist of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques.

Preoperative procedures:

Patients who have inadequate crown length and width ratio or short clinical crown will receive esthetic crown lengthening procedure to adjust gingival levels before being included in this study.

Clinical photographs:

Clinical photographs will be taken at baseline, 2 weeks, 1 month, 3 months postoperatively.

Intervention group I:

Patients in the intervention group I will take zinc gluconate 50 mg (Now food company) 1 per day to increase zinc level with phytase supplement 176mg (800FTU) (Goodphyte company) 2 tablets per day to give the maximum absorption of zinc, both supplements will be given for 4 days before botulinum toxin injections.

Intervention group II:

Patients in the intervention group II will take zinc gluconate 50 mg (Now food company) 1 per day to increase zinc level, 4 days before botulinum toxin injections.

Control group:

Patients in the control group will receive the Botulinum toxin injections only.

Botulinum toxin type A injection:

The patients will be injected at both sides into the "Yonsei point," (3Units) the point that would target 3 muscles responsible for upper lip elevation during smiling, including the levator labii superioris alaeque nasi (LLSAN), in a single injection. This landmark will be identified as the center of a triangle formed by the convergence of the LLSAN, the levator labii superioris (LLS), and the Zygomaticus minor muscles and is located 1 cm lateral to the ala horizontally and 3 cm above the lip line vertically in both men and women (Hwang et al. 2009) and (Nasr et al. 2015).

Postoperative care:

After Botox injection the patients will be instructed to:

1. Remain upright for 4 hours after injection (patients may lie in a reclined position, but not lay flat)
2. Refrain from aerobic exercise that increases the heart rate.
3. Not to massage or manipulate injected areas for 24 hours after injections,
4. Refrain from using ibuprofen, for 24 hours following injection.
5. If bruising appears, apply ice to area for 15 minutes every hour to decrease bruising.

Follow up:

Botox will gradually take effect over 7-10 days with optimum result at 2 weeks. After 2 weeks the patients would come for an additional touch up dose (1 unit at each injection point)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with excessive gingival display >3mm and with normal clinical crown dimensions.
2. Adults >18 years.
3. Non-smokers.
4. Systemically healthy.
5. Hypermobile lip and mild VME.

Exclusion Criteria:

1. Severe VME.
2. Pregnant or lactating females.
3. Patients with inflamed gingiva or gingival enlargement.
4. Inflammation or infection at the site of injection.
5. Patients with known allergy to any of the components of BTX-A or BTX-B (i.e. BTX, human albumin, saline, lactose and sodium succinate).
6. Patients using anticholinesterase or other agents interfering with neuromuscular transmission.
7. Psychologically unstable or who have questionable motives and unrealistic expectations.
8. Dependent on intact facial movements and expressions for their livelihood (e.g. actors, singers, musicians and other media personalities).
9. Afflicted with a neuromuscular disorder (e.g. myasthenia gravis, Eaton- Lambert syndrome).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Gingival display | The gingival display will be measured at baseline, 2 weeks, 4 weeks, 2 months, 3 months.
  To measure the amount of gingival display, a digital camera will be used to take the close up perioral as well as frontal smiling photographs. Care will be taken to capture a nonposed spontaneous smile. A measuring scale with ruler will be used for standardization of the photographs.

SECONDARY OUTCOMES:
Patient satisfaction (smile self-assessment) | 2 weeks, 3 months
  Will be measured by using questionnaire using Likert scale
  1. Very dissatisfied
  2. Dissatisfied
  3. Neutral
  4. Satisfied
  5. Very satisfied
Electrical activity of the smile muscles (EMG) | baseline, 2 weeks and 3 months
  The compound muscle action potential is an electromyography investigation that measures the simultaneous action potentials for a group of muscle fibers in the same area
Smile type | baseline, 2 weeks and 3 months:
  Classification by (Rubin 1974) according to neuromuscular smile pattern
  Three main types:
  The commissure smile: Mona Lisa smile, where the corners of the mouth are pulled up and outward followed by the levators of the upper lips contracting to show the upper teeth.
  The cuspid (canine) smile: The levator labii superioris are dominant. They contract first, exposing the canine teeth. The corners of the mouth contract secondarily to pull the lips upward and outward.
  The complex smile: all the elevators of the lips, the elevators of the corners of the mouth, and the depressors of the lower lips contract at the same time to show all the upper and lower teeth
Esthetics (Symmetry) for operators | baseline, 2 weeks and 3 months:
  A group of 12 dentists will evaluate the before and after photographic records and rate the results on a 1 to 5 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Weam A El-Battawy, Ass. Prof., Study Director — Cairo University; Mawda M Hussain, Bachelor, Principal Investigator — Cairo University; Nesma F Shemais, lecturer, Study Chair — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt